CLINICAL TRIAL: NCT03546088
Title: Awake Nasal Intubation With a Flexible Nasolaryngoscope in Patients With Laryngeal, Oro and Hypo-pharynx Tumours With Midazolam-fentanyl-droperidol Sedation Protocol- Technique and Patient Satisfaction
Brief Title: Awake Nasal Intubation in Laryngopharyngeal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Marchis Ioan Florin, Principal Investigator- Head of the Anaesthesia Dept. of ENT Clinic- Cluj Napoca, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: marchisioan
Record Dates: First submitted 2018-05-01; First posted 2018-06-06 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Airway Management
Keywords: awake intubation; nasal fiberscope; topical anesthesia
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- awake naso-tracheal intubation (Experimental): The patients with obstructive oro and hypo-pharynx tumours will have their airway secured through awake fiberoptic naso-tracheal intubation with light sedation and topical anaesthesia with lidocaine. The sedation will be provided in small boluses until the desired level will be achieved not exceeding 0.05 mg/kg of midazolam and 3 mcg/kg fentanyl. The dose of lidocaine will be to a maximum of 7 mg/kg. The reinforced intubating tube will be lubricated with lidocaine gel.
  Interventions: Device: fiberoptic naso-tracheal intubation; Drug: Topical anaesthesia; Drug: Light sedation

INTERVENTIONS:
Device: fiberoptic naso-tracheal intubation — The trachea will be intubated under direct fiberoptic view after a fiberoptic upper airway examination. The flexible nasolaryngoscope will be armed with an intubating tube and passed inside tracheal lumen trough one of the nostrils.
Drug: Topical anaesthesia — Topical anaesthesia with lidocaine will be provided through nebulisation and instillation. The intubating tube will be lubricated with a gel containing lidocaine.
Drug: Light sedation — The patient will be sedated with a combination of midazolam, fentanyl administered intravenously in small boluses until the desired level of sedation is achieved as expressed of The Observer's Assessment of Alertness/Sedation Scale (OAA/S) of 4 or 5.

SUMMARY:
This study evaluates the efficiency of awake naso-tracheal intubation and patient satisfaction when using a small diameter flexible nasolaryngoscope together with topical anaesthesia and light sedation with a combination of benzodiazepine and fentanyl. The selected patients will have difficult airway access because of obstructing oro- and hypo-pharynx tumours.

DETAILED DESCRIPTION:
Awake naso-tracheal fiberoptic intubation is an established method of securing a difficult airway. The patient's comfort and optimum intubation conditions are paramount for success. The study proposes to analyse a series of patients with obstructive pharyngo-laryngeal pathology, following the degree of satisfaction, reliability of the procedure and any incidents or complications.

Awake intubation could be the safest way to control difficult airway as the patient maintains spontaneous respiration and intact reflexes. Main concerns for the success of this procedure should be a good technique, a calm and cooperative patient and good preparation with careful topical anaesthesia and appropriate sedation. The tool used in this study will be a flexible nasolaryngoscope of 2.9 mm diameter and 300 mm working length which might offer an advantage over lengthier fiberscopes in matter of manoeuvrability and patient comfort. Prior intubation the patients will have an upper airway fiberscopic exam from nostrils to tracheae with the same tool.

ELIGIBILITY:
Inclusion Criteria:

* patients with tumours of larynx, oro and hypo-pharynx that obstruct airway access.

Exclusion Criteria:

* Patients who refuse the procedure, with bleeding disorders, acute respiratory failure manifested by stridor or the impossibility of nasal passage are excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
The duration of the procedure | 10 minutes
  The duration of the successful naso-tracheal intubation, starting from the passage of the intubating tube through one of the nostrils until the endotracheal intubation confirmation by free bag movement and capnography.

SECONDARY OUTCOMES:
Momentary discomfort shown by coughing, grimacing, constricting vocal cords, limb movement or blunt cardiovascular response | 10 minutes
  Expressed by grimacing, coughing , laryngospasm or constricting vocal cords, limb movement, a cardiovascular response of more than 20% variation in mean arterial pressure or cardiac frequency, rhythm disturbances.
Early and late complications | During procedure and 48 hours post-procedure
  monitoring incidents which could appear during or after the procedure (failure of achieving tracheal intubation, respiratory or cardio-vascular life threatening incidents, local injuries, bleeding, accidental tube displacement or blocking)
Patient satisfaction about the procedure at 24 hours post-procedure | 24 hours
  The subjects will complete a satisfaction questionnaire, in the form of a visual analogue scale. The scale will have the form of a 10 cm line marked with five grades of their discomfort during the procedure: none, mild, moderate, very bad and unbearable. Above this written words there is a 1 to 10 scale on which the patient will note there satisfaction score- 1 is the corespondent of no discomfort and 10 is for unbearable. The patient will fill in the scale the day after surgery. An average of the score of all patients will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Ioan Florin Marchis, Md, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy
Locations (1):
- Cluj County Emergency Hospital- ENT Clinic, Cluj-Napoca, Cluj, Romania